CLINICAL TRIAL: NCT00890344
Title: "Body Composition Assessment in Healthy Full-term Neonates by Anthropometry, Air Displacement Plethysmography (PeaPod) and Multiple-frequency Bio-impedance Analysis (BIA)"
Brief Title: Body Composition Assessment in Healthy Full-term Neonates by Anthropometry, Air Displacement Plethysmography and Multiple-frequency Bio-impedance Analysis
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Annes Omnes, University Hospital of Nantes
Other Study IDs: BRD08/7-P
Record Dates: First submitted 2009-04-27; First posted 2009-04-29 (Estimated); Last update posted 2011-09-30 (Estimated); Status verified 2011-09

CONDITIONS: Neonates
Keywords: PeaPod; BIA; Anthropometry; Body Composition; Fat Mass; Total Body Water; Neonatology

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Low birth weight and prematurity are associated with adverse metabolic outcome in adult life. Yet it remains to be determined whether this outcome is the consequence of the low birth weight per se, or of the catch up growth achieved in Neonatology units using an early, 'aggressive' nutritional management. As a matter of fact, 'aggressive' nutrition may promote fat mass, rather than lean body mass accretion. Assessment of body composition therefore is key to evaluate the efficacy of the nutritional management of these infants. Scarce data is, however, available in the literature about the body composition of healthy full-term neonates in the first few days of life.

The aim of this study is to:

1. Evaluate the feasibility and reproducibility of a safe and non invasive method of measurement of infant body composition by Air Displacement Plethysmography (PeaPod). Anthropometry and BIA will be used as the reference techniques to assess the accuracy of the PeaPod
2. Describe the body composition (fat mass, fat free mass) of healthy full-term neonates in the first few weeks of life
3. Obtain data on the total body water content of healthy full term infants from BIA.

ELIGIBILITY:
Inclusion Criteria:

* Full-term infants
* 10th percentile for gestational age, according to the Audipog's growth chart

Exclusion Criteria:

* Congenital diseases
* Chromosomal abnormalities
* Any disease requiring intensive care

Max Age: 1 Day | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Full-term infants 10th percentile for gestational age, according to the Audipog's growth chart
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2009-02; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Accuracy and reproducibility of the PeaPod compared with Anthropometry and BIA. We defined that assessments are convergent if the difference between methods is less than 10 percent. | August 2009

SECONDARY OUTCOMES:
Describe the body composition (fat mass, fat free mass) of healthy full-term neonates To get data on the total body water that we can refer to from BIA. | August 2009

CONTACTS AND LOCATIONS:
Overall Officials: Anne CA FRONDAS-CHAUTY, Dr, Principal Investigator — Nantes University Hospital
Locations (1):
- Centre Hospitalier Universitaire, Nantes, France